CLINICAL TRIAL: NCT05962996
Title: Evaluation of Pain Levels by Quantitative Pupillometry During the Placement of Deep Venous Catheters in Sedated Patients in Intensive Care Unit
Brief Title: Evaluation of Pain Levels by Quantitative Pupillometry During the Placement of Deep Venous Catheters in Sedated Patients in Intensive Care Unit (PUPICAT)
Acronym: PUPICAT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Universitaire de Tours (Other Government)
Collaborators: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Principal Investigator, Ambre Sauvage, Principal Investigator, Centre Hospitalier Régional Universitaire de Tours
Other Study IDs: DR230092; 2023-A00712-43 (Other: IdRCB)
Record Dates: First submitted 2023-06-22; First posted 2023-07-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness
Keywords: Pupillometry
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amines: Sedated and intubated patients requiring a deep venous catheter, unable to communicate their level of pain, and treated with aminergic drugs (no curare) Assessment of pain levels by pupillometry during the placement of the deep venous catheter
  Interventions: Device: Pupillometry
- Curares: Sedated and intubated patients requiring a deep venous catheter, unable to communicate their level of pain, and treated with curares (no aminergic drug) Assessment of pain levels by pupillometry during the placement of the deep venous catheter
  Interventions: Device: Pupillometry
- Sedation alone: Sedated and intubated patients requiring a deep venous catheter, unable to communicate their level of pain, without any aminergic drug nor curare Assessment of pain levels by pupillometry during the placement of the deep venous catheter
  Interventions: Device: Pupillometry

INTERVENTIONS:
Device: Pupillometry — Measurement of pain levels by pupillometry during the insertion of a deep venous catheter

SUMMARY:
Pain is common in intensive care and gives rise to multiple consequences that can impact the future of patients. The placement of deep venous catheters are painful gestures of common practice in intensive care. However, some patients are ventilated and sedated and their level of pain is difficult to judge. Quantitative pupillometry seems to be a reliable tool for assessing pain in these patients unable to communicate. The method is already common practice in the operating room for this indication and recent studies increasingly validate its use in intensive care.

The aim of the study is to validate the different levels of pain that can be assessed by pupillometry within this population during catheterization and to identify any non-responding subgroups (in order to conduct future clinical trials evaluating pain therapies).

DETAILED DESCRIPTION:
Three groups of patients will be studied : with aminergic drugs / with curare / without aminergic drugs nor curare.

The measurement of pain levels by quantitative pupillometry (NPi®-200 pupillometer, NeurOptics® USA) will be made in intubated, sedated patients, unable to communicate on their level of pain during the placement of a deep venous catheter.

Pain will be evaluated before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter.

Simultaneously, RASS and BPS scores as well as the patient's vital parameters and the cumulative doses of sedation-analgesia, curare and aminergic drugs will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 hospitalized in Intensive Care Unit
* Requiring the placement of a deep venous catheter (central venous catheter or dialysis catheter)
* Sedated, intubated, unable to communicate about pain
* No opposition to participation in the study

Exclusion Criteria:

* Any ophthalmological pathology (lesion of the orbital cavity, edematous soft tissue or with an open lesion)
* Any intracranial pathology (stroke, subarachnoid hemorrhage, tumour, etc.)
* Patient post-cardio-respiratory arrest within the first 48 hours
* Medicines interfering with the pupillary reflex: clonidine dexmedetomidine, droperidol, metoclopramide, nitric oxide, scopolamine, atropine
* Patient protected within the law
* Previous participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU, sedated, intubated, unable to communicate their levels of pain and requiring the placement of a deep venous catheter
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in variation of pupillary diameter by quantitative pupillometry | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Pupillary variation (%) = [maximum pupil diameter (mm) - minimum pupil diameter (mm)] / maximum pupil diameter (mm)]

SECONDARY OUTCOMES:
Changes in pupillary reflex latency by quantitative pupillometry | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Latency of pupillary reflex in seconds
Changes in pupil constriction by quantitative pupillometry | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Pupil constriction speed in mm/s
Changes in pupil dilatation by quantitative pupillometry | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Pupil dilation speed in mm/s
Changes in NPi by quantitative pupillometry | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Neurological Pupil Index (NPi), from 0 to 4.9, higher scores meaning a better outcome (normal pupillary light reflex)
Changes in BPS scores | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Behavioural Pain Scale scores : from 3 to 12, higher scores meaning a worse outcome (more pain)
Changes in respiratory rate | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Respiratory rate (cycles per minute)
Changes in heart rate | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Heart rate (beats per minute)
Changes in blood pressure | During the insertion of the deep venous catheter : before starting the placement of the catheter, at puncture(s), at dilation(s), and during the suture of the catheter (through study completion : an average of 20 minutes)
  Blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU d'Orléans, Orléans
  - CHRU de Tours, Tours